CLINICAL TRIAL: NCT00812084
Title: Collecting Health Outcomes and Economic Data on Hospitalized Community-Acquired Pneumonia - a Prospective Cohort Study
Brief Title: Costs, Health Status and Outcomes of CAP (Community-Acquired Pneumonia)
Acronym: CHO-CAP
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, G.A. de Wit, PhD, MSc, UMC Utrecht
Other Study IDs: 6115A1-3015
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Pneumonia
Keywords: Quality of life; health resources; costs; community-acquired pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CAP cohort: Includes cases that were hospitalized because of a community-acquired pneumonia during the study period, and for which we had a baseline EQ-5D score from the start of the study period. These CAP cases are prospectively followed for up to one year using questionnaires for health status and (health) resources.
- Controls cohort: For each CAP cases, two controls are matched based on age, sex and baseline EQ-5D score measured at the start of the study. These controls are prospectively followed for up to one year using questionnaires for health status and (health) resources.

SUMMARY:
The purpose of this study is to collect additional data on hospitalized Community-Acquired Pneumonia (CAP) on health states, health outcomes and on (health) resources and estimate the differences in the quality of life and resources of elderly persons with and without CAP.

DETAILED DESCRIPTION:
Within the study data on quality of life and various health and non-health resources and their costs is collected with the help of questionnaires administered at different points in time in different cohorts. Data collection is additional upon data collected in the main CAPITA trial, such as incidence data, mortality estimates, use of some health care resources, vaccine effectiveness and general background (socio-demographic) data.

In a first sub-study of CHO-CAP, the CAPITA participants are asked, via written information distributed shortly after vaccination, to fill in once-only a short questionnaire describing their health status (5 item EQ-5D instrument) and a few additional socio-demographic background data. This is done in order to determine an EQ-5D baseline score (index value for health status) - a prerequisite to match CAP patients and controls later, and as such an inclusion criterion for the two (nested) cohorts that will be followed prospectively.

About 2,000 cases of CAP are expected to occur in the CAPITA cohort in the next two to three years. Assuming a response rate of ~30% for the baseline questionnaire, we will have some 600 CAP cases out of the 2,000 expected patients for whom a baseline EQ-5D score is available. These CAP patients will be asked to participate in a prospective cohort study. Within CHO-CAP, these CAP cases will be followed for up to one year after their CAP episode. For each CAP case included in the CAP cohort, two controls from the baseline population are matched and included in a cohort of controls (non-CAP elderly with similar baseline health status). Controls will also be followed for up to one year. The matches between CAP cases and controls will be made based on age, sex and EQ-5D baseline score. This implies that controls will only be recruited from the group that responded to the baseline measurement of health status shortly after vaccination. For both cohorts, the CAP patients and the matched controls, additional data on health care and non-health care resource use, on health status, using EQ-5D and SF-36 questionnaires, and on selected health outcomes is collected at four contact (at 0, 1, 6 and 12 months) moments within a period of 1 year. This will be done using questionnaires, distributed during a home visit and by post.

ELIGIBILITY:
Inclusion Criteria:

* Only participants of the CAPITA trial. Therefore the inclusion criteria as applied in CAPITA are the baseline for the current study. Additionally all participants had to be consent and had to fill in a baseline EQ-5D questionnaire
* Additionally for CAP patients: Consent to be filling to participate as a CAP and the presence of CAP has to be confirmed by the independent adjudication committee of the main CAPITA trial
* Additionally for controls: Consent to be filling to participate as control

Exclusion Criteria:

* The non-availability of a baseline EQ-5D score is an exclusion criterion for the prospectively followed cohorts (both CAP patients and controls)
* In all stages of the study, patients have the right to withdraw their consent and stop their participation in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of community-dwelling persons 65 years and older and taking part in the CAPITA trial, in total 85,000 persons
Sampling Method: Non-Probability Sample
Enrollment: 48634 (Actual)
Dates: Start 2008-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
(Differences in) the quality of life/health status of elderly persons with and without CAP; inclusive of a 12-months follow-up period after occurrence of a CAP | 12-months follow-up after CAP
(Differences in) the resources use (health care and non-health care) by CAP patients and non-diseased controls; inclusive of follow-up of 12 months after discharge | 12-months follow-up after CAP

SECONDARY OUTCOMES:
To describe the baseline health status and quality of life in a community-dwelling population of 65 years and older | at the begin of the study

CONTACTS AND LOCATIONS:
Overall Officials: G.Ardine de Wit, PhD, Principal Investigator — Julius Center for Health Sciences and Primary Care; UMC Utrecht; Marc J.M. Bonten, Prof., MD PhD, Principal Investigator — Julius Center for Health Sciences and Primary Care; UMC Utrecht
Locations (1):
- Questionnaires are filled in at participants home addresses, The Netherlands, Netherlands

REFERENCES:
- [Derived] Mangen MJ, Huijts SM, Bonten MJ, de Wit GA. The impact of community-acquired pneumonia on the health-related quality-of-life in elderly. BMC Infect Dis. 2017 Mar 14;17(1):208. doi: 10.1186/s12879-017-2302-3. PMID 28292280
- [Derived] Mangen MJ, Bolkenbaas M, Huijts SM, van Werkhoven CH, Bonten MJ, de Wit GA. Quality of life in community-dwelling Dutch elderly measured by EQ-5D-3L. Health Qual Life Outcomes. 2017 Jan 6;15(1):3. doi: 10.1186/s12955-016-0577-5. PMID 28069062
- [Derived] Mangen MJ, Bonten MJ, de Wit GA. Rationale and design of the costs, health status and outcomes in community-acquired pneumonia (CHO-CAP) study in elderly persons hospitalized with CAP. BMC Infect Dis. 2013 Dec 19;13:597. doi: 10.1186/1471-2334-13-597. PMID 24354588
- See also: The CHO-CAP study uses the CAPITA research infrastructure to collect additional data on hospitalized CAP not covered in the main trial. CAPITA is registered with clinicalTrials.gov as: NCT00744263. — http://www.clinicaltrials.gov/ct2/show/NCT00744263?term=pneumonia+AND+netherlands&rank=6